CLINICAL TRIAL: NCT05529303
Title: The Effect of the "Feminine Identity Improvement Program" Based on Cognitive Behavioral and Expressive Techniques Applied to Gynecological Cancer Patients on Prolonged Grief Reactions and the "Perception of Femininity"
Brief Title: Prolonged Grief and Perception of Femininity in Gynecological Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kevser Pamuk (Other)
Responsible Party: Sponsor-Investigator, Kevser Pamuk, Instructor, Afyonkarahisar Health Sciences University
Organization: Afyonkarahisar Health Sciences University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AfyonkarahisarHSU-KPAMUK-1
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Cervix Cancer; Uterine Cancer; Ovarian Cancer; Endometrial Cancer; Vulva Cancer; Grief; Femininity
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Vulvar Neoplasms; Femininity | interventions — Art Therapy; Play Therapy

STUDY DESIGN:
Intervention Model Description: The Prolonged Grief Disorder-Patient Form will be administered to all gynecological cancer patients who meet the inclusion criteria. The patients with the highest prolonged grief reaction as much as the number of samples determined will be included in the study by dividing them into groups through block randomization.
Who Masked: Outcomes Assessor
Masking Description: The evaluation of the data will be carried out by an independent researcher who will be blinded to the intervention and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group determined by the randomization method will be given the 'Feminine Identity Improvement Program', based on cognitive behavioral and expressive techniques, which is structured to be 90-120 minutes once a week for 10 weeks. The program to be applied to the intervention group has been created by the researcher in line with the literature review and the necessary expert opinions were obtained.
  Interventions: Behavioral: Such as art therapy, play therapy, breathing techniques
- Control group (No Intervention): No intervention will be applied to the control group during the study.

INTERVENTIONS:
Behavioral: Such as art therapy, play therapy, breathing techniques — The Cognitive Behavioral Therapy (CBT) model suggests that the individual's dysfunctional thoughts about self, the world, and/or others are based on irrational or illogical assumptions. An individual's self and his/her view of the world are central to the determination of his/her feelings and behaviors and thus can be changed through changing the individual's thoughts, feelings, and behaviors. CBT techniques are in line with the use of expressive art techniques. The common goal in both CBT and expressive arts is to achieve behavior change in the individual. An intervention program has been prepared by the researcher in line with this literature information.
  Arms: Intervention group

SUMMARY:
The aim of this study is to determine the effect of the 'Feminine Identity Improvement Program', based on cognitive behavioral and expressive techniques applied to gynecological cancer patients, on prolonged grief reactions and the perception of femininity. The study will be conducted in a randomized controlled and qualitative type with gynecological cancer patients who completed their surgical treatment at least three months ago in the last year at Afyonkarahisar Health Sciences University Hospital.

DETAILED DESCRIPTION:
The Personal Information Form and the Prolonged Grief Disorder Scale will be used as data collection tools in the study. The Prolonged Grief Disorder Scale-Patient Form will be applied to all gynecological cancer patients who meet the inclusion criteria for the study. When the literature was examined for the planned study, we could not come across any study that used the scale to be applied or a parallel form of it. Since it will be a reliable method to perform power analysis with the values obtained by conducting a pilot study in the absence of literature reference, the power analysis process will be performed by carrying out a pilot study with a total of 30 cases. The study will be terminated if a sample number is determined to be 30 or fewer as a result of the power analysis. If the sample number exceeds 30, the number of samples will be increased as much as the difference. Accordingly, the patients with the highest prolonged grief reaction as much as the number of samples determined will be included in the study by dividing them into groups through block randomization. The intervention group determined by the randomization method will be given the 'Feminine Identity Improvement Program', based on cognitive behavioral and expressive techniques, which is structured to be 90-120 minutes once a week for 10 weeks. The program to be applied to the intervention group has been created by the researcher in line with the literature review and the necessary expert opinions were obtained. No intervention will be applied to the control group during the study. In order to determine the effect of the program, measurements will be carried out in both groups before the program (pre-test), at the end of the program (post-test-10th week), and three (3) months after the end of the program. In order to evaluate the perception of femininity, individual interviews will be conducted at the end of the program with the intervention group patients until saturation is reached. Since no scale evaluates the perception of femininity in the literature, the perceptions of femininity will be evaluated with individual interviews accompanied by the guide interview form prepared by the researchers in line with the literature. After the completion of the study, the program will be repeated with the volunteers from the control group.

ELIGIBILITY:
Inclusion Criteria:

* To be in the age range of 18-65 years,
* To have been diagnosed with gynecological cancer,
* To be aware of the diagnosis of cancer,
* At least 3 (three) months have passed after the completion of the surgical treatment
* To be able to read and write
* Voluntary participation in the study.

Exclusion Criteria:

* Having a diagnosis of any psychiatric disorder
* Having any disability (physical, mental, vision, hearing, speaking..)
* Being in terminal phase.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-02-26 (Actual); Primary Completion 2023-05-07 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Prolonged Grief Disorder Score | Before determining the intervention and control group
  The scale used to evaluate the emotional experiences and grief reactions of cancer patients regarding the loss caused by the disease was scored on a Likert-type scale (1=never, 5=many times a day for items 1-4.;1=never, 5=too many for items 5-12.) There are 12 items.
  An increase in the total score obtained from the scale indicates an increase in grief symptoms.
Prolonged Grief Disorder Score | At the end of the intervention program (week 10)
  The scale used to evaluate the emotional experiences and grief reactions of cancer patients regarding the loss caused by the disease was scored on a Likert-type scale (1=never, 5=many times a day for items 1-4.;1=never, 5=too many for items 5-12.) There are 12 items.
  An increase in the total score obtained from the scale indicates an increase in grief symptoms.
Prolonged Grief Disorder Score | 3 months after the end of the intervention program (5.5 months)
  The scale used to evaluate the emotional experiences and grief reactions of cancer patients regarding the loss caused by the disease was scored on a Likert-type scale (1=never, 5=many times a day for items 1-4.;1=never, 5=too many for items 5-12.) There are 12 items.
  An increase in the total score obtained from the scale indicates an increase in grief symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Karaca, Study Director — Duzce University
Locations (1):
- Kevser Pamuk, Merkez, Afyonkarahisar, Turkey (Türkiye)